CLINICAL TRIAL: NCT05224492
Title: Sulforaphane Use to Effect Inflammatory and Metabolic Changes in Virally Suppressed HIV Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Specialty Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSHC1001
Record Dates: First submitted 2022-02-01; First posted 2022-02-04 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane Group (Experimental)
  Interventions: Drug: Sulforaphane
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sulforaphane — 40 mg of Sulforaphane powder once daily.
  Arms: Sulforaphane Group
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Assess the effects of Sulforaphane supplementation in HIV patients that have achieved viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients on active treatment who have a suppressed viral load and have been virally suppressed for 6 months or more.
* BMI increase of 10% or more since initiation of HIV treatment over a year period.
* BMI equal to or greater than 30.
* 18-85 years of age.

Exclusion Criteria:

* Cancer
* Pregnancy or breastfeeding
* Intolerance to cruciferous vegetables
* Intolerance to sulforaphane
* Gluten Intolerance
* Creatinine > 1.3 mg/dL
* GFR < 60
* AST or ALT > 1.5 times upper limit of normal.
* White cell count < 2000 cells per ml.
* Hemoglobin < 10.5 g/dL.
* Platelet count < 140,000 per ml.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-21 (Estimated); Primary Completion 2022-07-21 (Estimated); Study Completion 2022-09-21 (Estimated)

PRIMARY OUTCOMES:
Lipids | 4 months
  Triglycerides, Cholesterol
Inflammatory Markers | 4 months
  CRP

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Giron, MD, Principal Investigator — Sunshine Specialty Health Care

IPD SHARING:
Plan to Share IPD: Undecided